CLINICAL TRIAL: NCT02172170
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (0.5 mg to 800 mg) of BI 10773 as Tablets Administered to Healthy Male Subjects. A Randomised Placebo-controlled (Within-dose Groups) and Double-blind Trial.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 10773 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.1
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- BI 10773 single rising dose (Experimental)
  Interventions: Drug: BI 10773 single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 10773 single rising dose
  Arms: BI 10773 single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of single rising oral doses of BI 10773 to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs ((blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age ≥ 18 and Age ≤ 50 years
3. BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination including ((blood pressure (BP), pulse rate (PR), 12-lead electrocardiogram (ECG)) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with the dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms);
21. A history of additional risk factors for torsade de pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome);

    Exclusion criteria specific for this study:
22. Elevated urinary glucose levels at screening (> 15 mg/dl; > 0.83 mmol/L)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 33 days
Number of patients with clinically significant changes in vital signs | up to 12 days
Assessment of tolerability by investigator on a 4-point scale | up to day 4
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 12 days
Number of patients with abnormal findings in physical examination | up to 12 days
Number of patients with abnormal changes in laboratory parameters | up to 12 days

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
λz (terminal rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 72 hours after drug administration
CL/F (total clearance of the analyte in the plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Ae t1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 72 hours after drug administration
fe t1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 72 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 72 hours after drug administration